CLINICAL TRIAL: NCT06014684
Title: Timing Exercise Training as Strategy to Improve Insulin Sensitivity and Substrate Metabolism in Men and Woman With Pre-diabetes
Acronym: Timed Training
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NL83421.068.22
Record Dates: First submitted 2023-07-20; First posted 2023-08-28 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Pre-diabetes; Overweight and Obesity
MeSH Terms: conditions — Glucose Intolerance; Overweight; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- AM exercise (Experimental): HIIT program performed between 07:00-09:00 AM
  Interventions: Behavioral: Timing of exercise
- PM exercise (Experimental): HIIT program performed between 15:00-17:00 PM
  Interventions: Behavioral: Timing of exercise

INTERVENTIONS:
Behavioral: Timing of exercise — High Intensity Interval Training (HIIT) program for 12 weeks (3 per week/36 sessions in total)

SUMMARY:
n a retrospective analysis of an exercise training program performed either in the morning or afternoon, we found that the afternoon training group improved their peripheral insulin sensitivity and fasting plasma glucose levels to a greater extent than the morning group. However, underlying mechanisms are unclear.

The primary study endpoint is nocturnal glucose levels measured by a continuous glucose monitor (CGM).

DETAILED DESCRIPTION:
Rationale: Various metabolic processes, including resting metabolic rate, insulin sensitivity and insulin secretion, follow a recurring 24-hour cycle. These rhythms are shown to be disturbed in in pre-diabetes volunteers compared to young healthy volunteers. In a retrospective analysis of an exercise training program performed either in the morning or afternoon, we found that the afternoon training group improved their peripheral insulin sensitivity and fasting plasma glucose levels to a greater extent than the morning group. However, underlying mechanisms are unclear.

Objective: The main objective of this study is to determine whether prolonged exercise training in the afternoon (15:00-17:00 PM) differs from exercise training in the morning (07:00-09:00 AM) in improving insulin sensitivity in individuals with pre-diabetes, and to investigate its underlying mechanisms.

Study design: The present study is a randomized double arm longitudinal intervention study in a pre and post design.

Study population: 24 pre-diabetic individuals (men and postmenopausal women aged 40 - 75 years and with BMI ≥ 25 and ≤ 38 kg/m2) will complete this study (12 participants in the morning training group and 12 participants in the afternoon training group). From experience with similar studies, we estimate a drop-out rate of 20% and a screening failure of 70% (because individuals often do not know they are pre-diabetic). This results in maximally 30 participants that have to be included and 100 participants that have to be screened (maximally).

Intervention (if applicable): Participants will perform a 12-weeks supervised high intensity interval training (HIIT) program with three ~30 min exercise sessions per week. Participants will be randomly assigned to the morning or afternoon training time. To assess the outcomes, participants will come to the university for a 43h measurement period both before and after the 12-week training program.

Main study parameters/endpoints: The primary study endpoint is nocturnal glucose levels measured by a continuous glucose monitor (CGM). The secondary outcomes are 24h energy and substrate metabolism. Exploratory outcomes are body composition, intrahepatic lipid content and composition, hepatic insulin sensitivity, hepatic glycogen levels, maximal aerobic capacity, skeletal muscle oxidative capacity, visceral and subcutaneous adipose tissue volume, sleeping metabolic rate, blood glucose levels (continuously measured over 7days) and immune responses.

ELIGIBILITY:
Inclusion Criteria:

* Aged 40-75 years.
* Body mass index (BMI) ≥25 kg/m2
* Male, or postmenopausal (at least 1 year post cessation of menses) female
* Pre-diabetes based on one or a combination of the following criteria:

  * Impaired Glucose Tolerance (IGT): plasma glucose values ≥ 7.8 mmol/l and ≤ 11.1 mmol/l 120 minutes after glucose drink consumption during OGTT in screening
  * ImpairedFastingGlucose(IFG):Fastingplasmaglucose≥6.1mmol/land≤6.9 mmol/l
  * Insulin Resistance: glucose clearance rate ≤ 360 mL/kg/min, as determined during the OGTT using OGIS120.
  * HbA1cof5.7-6.4%

Exclusion Criteria:

* Type 2 diabetes
* Patients with active congestive heart failure and and/or severe renal and or liver insufficiency
* Uncontrolled hypertension
* Any contra-indication for MRI scanning
* Alcohol consumption of >3 servings per day for man and >2 servings per day for woman
* Smoking
* Unstable body weight (weight gain or loss > 5kg in the last 3 months)
* Previous enrolment in a clinical study with an investigational product during the last 3 months or as judged by the Investigator which would possibly hamper our study results.
* Medication use known to hamper subject's safety during the study procedures.
* Subjects who do not want to be informed about unexpected medical findings.
* Men: Hb <8.0 mmol/L, Women: Hb <7.0 mmol/l
* Heavily varying sleep-wake rhythm (i.e. night shift work and travels across time zones).
* Significant food allergies/intolerance (seriously hampering study meals)
* Blood donation during or within 2 months prior to the study

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-07-13 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
nocturnal glucose levels | measured before and after the 12 weeks training program
  The main objective of this study is to determine whether prolonged exercise training in the afternoon differs from exercise training in the morning in improving nocturnal glucose levels insulin sensitivity in individuals with pre-diabetes.

SECONDARY OUTCOMES:
24h whole body energy expenditure | measured before and after the 12 weeks training program
  energy expenditure as measured by a 24h stay in the respiration chamber
24h substrate metabolism | measured before and after the 12 weeks training program
  24h substrate metabolism as measured by a 24h stay in the respiration chamber

OTHER OUTCOMES:
Body composition by Dual Energy X-ray Absorptiometry (DEXA) | measured before and after the 12 weeks training program
  fat-free mass (kg and percentage)
Body composition by Dual Energy X-ray Absorptiometry (DEXA) | measured before and after the 12 weeks training program
  fat mass (kg and percentage)
Intrahepatic lipid content and composition | measured before and after the 12 weeks training program
Hepatic glycogen levels | measured before and after the 12 weeks training program
VO2 max cycling test | measured before and after the 12 weeks training program
  measurement of participants' maximal aerobic capacity, absolute (L/min) and relative (ml/min/kg)
Skeletal muscle oxidative capacity | measured before and after the 12 weeks training program
  Ex vivo high-resolution respirometry using a two chamber Oxygraph (OROBOROS Instruments) will be performed. Multiple substrate/inhibitor titration protocols will be applied to extensively characterize the mitochondrial capacity of skeletal muscle fibers
Sleeping metabolic rate | measured before and after the 12 weeks training program
Blood glucose levels measured continuously over 7 days. | measured before and at the end the 12 weeks training program

CONTACTS AND LOCATIONS:
Locations (1):
- Maastricht University, Maastricht, Limburg, Netherlands